CLINICAL TRIAL: NCT00141180
Title: Placebo-Controlled, Randomized, Parallel Group, Multiple-Dose Study to Evaluate the Effects of CP-481,715 on Clinical Response and Cellular Infiltration Following Contact Allergen Challenge to the Skin of Nickel Allergic Subjects.
Brief Title: CP-481,715 Nickel Allergy Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3081018
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2005-11

CONDITIONS: Dermatitis, Allergic Contact
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — quinoxaline-2-carboxylic acid (4-carbamoyl-1-(3-fluorobenzyl)-2,7-dihydroxy-7-methyloctyl)amide

INTERVENTIONS:
Drug: CP-481,715

SUMMARY:
To evaluate the suitability of contact allergy as a method for the evaluation of c-chemokine receptor-1 antagonist.

ELIGIBILITY:
Inclusion Criteria:

* A history of nickel allergy confirmed by a visual positive reaction (graded at least ++) to T.R.U.E. TEST.

Exclusion Criteria:

* Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding contact allergic dermatitis or untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2003-09; Study Completion 2005-10

PRIMARY OUTCOMES:
Effect of CP-481,715 on clinical response and cell infiltration after nickel challenge

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (4):
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bryan, Texas
- Pfizer Investigational Site, Hellerup, Denmark